CLINICAL TRIAL: NCT03235843
Title: Rate Adaptive Atrial Pacing in Heart Failure Patients With Chronotropic Incompetence
Brief Title: Rate Adaptive Atrial Pacing in Heart Failure
Acronym: ADAPTION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: UMC Utrecht (Other); Maasstad Hospital (Other); Northwest Clinics Alkmaar (Unknown)
Responsible Party: Principal Investigator, Cornelis P. Allaart, Principal Investigator, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ISROTH20232
Record Dates: First submitted 2017-07-10; First posted 2017-08-01 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-08

CONDITIONS: Chronotropic Incompetence; Heart Failure; ICD
Keywords: Chronotropic Incompetence; Rate Adaptive Pacing; Minute Ventilation Sensor; Primary Prevention ICD Therapy; Implantable Cardioverter Defibrillator; Heart Failure; Exercise Intolerance
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Patients enter a double blind randomized cross-over pilot study and will be randomized in a 1:1 fashion to either rate responsive (MV sensor only) function on or off. After 3 months the pacing mode will be switched to the opposite mode.
Who Masked: Participant, Investigator
Masking Description: The pacing mode set by the pacemaker technician will not be disclosed to either patients or the study physician.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rate Adaptive Pacing ON (Active Comparator): AAIR pacing using a MV sensor
  Interventions: Device: AAIR pacing
- Rate Adaptive Pacing OFF (Placebo Comparator): DDI-pacing
  Interventions: Device: DDI-pacing

INTERVENTIONS:
Device: AAIR pacing — Rate adaptive pacing using a MV sensor.
  Arms: Rate Adaptive Pacing ON
Device: DDI-pacing — Rate adaptive pacing OFF
  Arms: Rate Adaptive Pacing OFF

SUMMARY:
The ADAPTION trial is an investigator initiated prospective randomized doubleblind cross-over pilot study in a multi-center setting.

Aim: to assess the ability of minute ventilation (MV) sensor driven rate adaptive atrial stimulation to restore functional capacity and quality of life in heart failure patients with chronotropic incompetence.

Methods: heart failure patients (left ventricular ejection fraction ≤35% & New York Heart Assessment II or III) who were implanted with a 2-chamber implantable cardioverter defibrillator (ICD) device equipped with a MV sensor that are diagnosed with chronotropic incompetence will be included in the study. Patients will be randomized in a 1:1 fashion to rate responsive pacing (MV sensor only) function ON (AAIR mode) or OFF (DDI mode). After 3 months the pacing mode will be switched to the opposite mode.

ELIGIBILITY:
Inclusion Criteria:

1. Chronotropic incompetence as assessed by a modified Heart Rate Score (mHRS)
2. Implanted with a Boston Scientific dual chamber ICD equipped with minute ventilation sensor
3. Symptomatic congestive heart failure (NYHA class II-III)
4. Left ventricular systolic dysfunction (LVEF <35%)
5. Optimal medical therapy
6. Sinus rhythm
7. Subjects should be able to perform normal daily activities

Exclusion Criteria:

1. Age <18 or incapacitated adult
2. Documented atrial fibrillation in the last 3 months prior to inclusion
3. Indication for pacing (SSS, AV conduction abnormalities requiring pacing)
4. Respiratory rate abnormalities (hyperventilation) or use of a mechanical ventilator
5. Patients who are unable to tolerate increased pacing rates
6. Indication for cardiac resynchronization therapy

Beta-blocker / ivabradine / amiodarone therapy is not an exclusion criterion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of quality of life | 3 months after changing the pacing mode
  Measured with the Minnesota Living with Heart Failure Questionnaire

SECONDARY OUTCOMES:
Improvement of functional capacity | 3 months after changing the pacing mode
  Measured with a six-minute walk test
Reversibility of chronotropic incompetence | 3 months after changing the pacing mode
  A comparison of the modified HeartRateScore with and without rate adaptive pacing.
Clinical status | 3 months after changing the pacing mode
  Measured with NYHA class assessment and number of hospitalizations for heart failure.
Daily activity level | 3 months after changing the pacing mode
  Measured with the device's accelerometer

CONTACTS AND LOCATIONS:
Overall Officials: Cornelis P Allaart, MD, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU university medical center, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brubaker PH, Kitzman DW. Chronotropic incompetence: causes, consequences, and management. Circulation. 2011 Mar 8;123(9):1010-20. doi: 10.1161/CIRCULATIONAHA.110.940577. No abstract available. PMID 21382903